CLINICAL TRIAL: NCT01622946
Title: The Effect of Topical Application of Tranexamic Acid in Total Hip Arthroplasty Through the Direct Anterior Approach. A Prospective, Double Blind, Placebo-controlled Clinical Trial.
Brief Title: The Effect of Topical Application of Tranexamic Acid in Total Hip Arthroplasty Through the Direct Anterior Approach
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2010-024410-59
Record Dates: First submitted 2012-06-14; First posted 2012-06-19 (Estimated); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Total Hip Arthroplasty; Postoperative Blood Loss
Keywords: total hip arthroplasty; tranexamic acid; postoperative blood loss
MeSH Terms: conditions — Postoperative Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Placebo (Active Comparator): The patients who receive placebo form the control group. The results can be compared with the results of the patients who did receive TXA
  Interventions: Drug: placebo
- Tranexamic acid (Placebo Comparator): The patients will receive 3g topical TXA for 15 minutes or 2 hours after THA. 33% of the patients will receive 3g of TXA trough a suction drain for 15 minutes after total hip arthroplasty, then the suction drain is opened. 33% will receive the same amount of TXA but the suction drain will only be opened 2 hours after application. The other patients will receive a placebo in the same manner
  Interventions: Drug: Tranexamic Acid

INTERVENTIONS:
Drug: Tranexamic Acid — 3g of tranexamic acid is topically applied after THA. The drugs is left for 15 minutes or 2 hours
  Arms: Tranexamic acid
Drug: placebo — The patients will receive 3g topical TXA for 15 minutes or 2 hours after THA. 33% of the patients will receive 3g of TXA trough a suction drain for 15 minutes after total hip arthroplasty, then the suction drain is opened. 33% will receive the same amount of TXA but the suction drain will only be opened 2 hours after application. The other patients will receive a placebo in the same manner
  Arms: Placebo

SUMMARY:
The effects of topical application of 3g tranexamic acid for 2 hours prior to opening of the suction drain following a total hip replacement

ELIGIBILITY:
Inclusion Criteria:

* patients who will receive a unilateral total hip arthroplasty

Exclusion Criteria:

* coagulopathy
* allergy to tranexamic acid
* preoperative anemia (a hemoglobin value of < 11g/dL in females and < 12g/dL in males)
* fibrinolytic disorders
* a history of arterial or venous thromboembolic disease
* pregnancy
* breastfeeding
* major comorbidities

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2020-04 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
postoperative blood loss in patients undergoing primary total hip arthroplasty | Haemoglobin levels, on which the postopererative blood loss is calculated, is measured preoperative and on day 1 and 4 postoperative

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Pellenberg, Pellenberg, Belgium